CLINICAL TRIAL: NCT03868891
Title: Device Assisted Exercises for Improving Soft Palate and Eustachian Tube Function in Children Between Ages 6-17 With or Without Cleft Palate and With Ventilation Tubes
Brief Title: Exercises for Improving Soft Palate and Eustachian Tube Function in Children With Ear Tubes With or Without Cleft Palate
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of funding
Sponsor: Noel Jabbour (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Noel Jabbour, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO18110061; 5R21DC017553-02 (NIH)
Record Dates: First submitted 2019-02-14; First posted 2019-03-11 (Actual); Results first posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-05

CONDITIONS: Cleft Palate; Tube Disorders Eustachian; Velopharyngeal Incompetence Due to Cleft Palate; Velopharyngeal Insufficiency
Keywords: Otitis media; Eustachian tube; Eustachian tube dysfunction; Eustachian tube function testing; Middle ear ventilation
MeSH Terms: conditions — Cleft Palate; Velopharyngeal Insufficiency; Otitis Media

STUDY DESIGN:
Intervention Model Description: experimental, open label
Masking Description: Researchers conducing Eustachian tube function testing and those conducing statistical analysis will be blinded to the visit number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- EMST150 (Experimental): Subjects with or without cleft palate will use the EMST150 2 times a day for 8 weeks.
  Interventions: Device: EMST150

INTERVENTIONS:
Device: EMST150 — The EMST150 consists of a handheld plastic tube with a mouthpiece on one end and an adjustable valve on the other end. Your child will close his/her lips around the mouthpiece and breathe out against resistance. The EMST150 will be adjusted to the point where airflow stops. Each day, your child will blow into the EMST150 5 sets of 5 times with a 10-15 second rest between each use and a 1-2 minute rest between each set of 5. You will adjust the resistance of the device each week, take a picture of the device settings, and document exercise sets performed in an exercise diary. These exercises will be performed twice in each nostril 2 times a day until your child's next visit at the MEPL (at least 8 weeks). Each session should take approximately 10-15 minutes, for a total of 30 minutes per day.
  Other Names: Expiratory Muscle Strength Trainer 150

SUMMARY:
Elevation of the soft palate (the soft part of the roof of the mouth) during swallowing helps the Eustachian tube to open and keep the ear healthy. (The Eustachian tube is the normal tube running from the middle ear to the back of the nose and throat). When the soft palate does not move enough (due to a history of cleft palate or for unknown reasons), this can lead to speech problems. Also, because the Eustachian tube is not opening enough, fluid can accumulate in the middle ear, which requires treatment with ear tubes. The goal of this research study is to determine if soft palate exercises will help improve the ability of the soft palate to close the area between the throat and nose, like it is supposed to during speech and swallowing, and if this improves Eustachian tube opening.

DETAILED DESCRIPTION:
This trial will look at the feasibility and effect of device-assisted soft palate exercises for the treatment of chronic Eustachian tube (ET) dysfunction (ETD) in older children still experiencing middle-ear disease. Children with or without cleft palate (CP) with ventilation tubes (VTs) will be evaluated for the function of the soft palate and the ET. Subjects with active muscular ETD and inadequate soft palate closure will be prescribed soft palate strengthening exercises for at least 2 months. The objective of the study is to demonstrate the effect of exercises on soft palate closure and ETF. This pilot study will enroll 30 children between ages 6-17 years with VTs or post-VT extrusion tympanic membrane (TM) perforations. All 30 children will have ETD, with active muscular dysfunction. 15 subjects will have a history of cleft palate (CP) and 15 no history of CP. Subjects will undergo history, physical examination including an ENT exam, video-otoscopy and ET function testing which may include Forced Response Test (FRT), Inflation-Deflation Test (IDT) and Tubomanometry. They will also undergo evaluations for swallow, speech and soft palate function. Enrolled children will then receive instruction on the use their EMST150 exercise device. This device will be used daily for at least 2 months. Subjects will undergo full evaluations for ET function and velopharyngeal incompetence after the 2-month treatment and will then discontinue the use of devices for at least 2 months. After this time, the same testing will be done. Weekly phone calls/emails/texts from study staff will encourage use of the devices as prescribed.

The following secondary outcome measures were part of the original study protocol but were eliminated after the start of the COVID-19 pandemic because the tests involved blowing maneuvers and risk of aerosolization. The protocol was modified to only include ETF tests that were necessary to achieve the goals of the study and that were safe for the participants.

'Velopharyngeal pressure after 2 months of exercise compared with baseline' 'Velopharyngeal pressure after 2 months of rest compared with baseline' 'Duration of velopharyngeal closure after 2 months of exercise compared with baseline' 'Duration of velopharyngeal closure after 2 months of rest compared with baseline' 'Ability to maintain velopharyngeal closure after 2 months of exercise compared with baseline' 'Ability to maintain velopharyngeal closure after 2 months of rest compared with baseline' 'Overall success in velopharyngeal closure after 2 months of exercise compared with baseline' 'Overall success in velopharyngeal closure following 2 months of rest compared with baseline'

The following other pre-specified outcome measures were removed for the same reason:

'Velopharyngeal pressure after 2 months of rest compared with pressure immediately following 2 months of exercise' 'Duration of velopharyngeal closure after 2 months of rest compared with pressure immediately following 2 months of exercise' 'Ability to maintain velopharyngeal closure after 2 months of rest compared with ability immediately following 2 months of exercise' 'Overall success in velopharyngeal closure following 2 months of rest compared with success immediately following 2 months of exercise'

'Eustachian tube function after 2 months of rest compared with function immediately following 2 months of exercise' was moved from an other pre-specified outcome measure to a secondary outcome measure due to its similar level of importance to the other secondary outcome measures.

Pressure chamber results were removed from outcome measures because they were unable to be obtained safely during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* 6-17 years old
* Otherwise healthy
* Currently have unilateral or bilateral ventilation tube(s) (VTs) inserted for otitis media with effusion (OME) or tympanic membrane retraction/retraction pocket (TM-R/RP) or a TM perforation after extrusion of a VT
* History of at least 2 sets of VT insertions in the past
* Eustachian tube (ET) function (ETF) tests showing an active muscular pattern of Eustachian tube dysfunction
* Some degree of velopharyngeal dysfunction during the ETF tests
* Cleft Palate (CP) cohort: non-syndromic; prior palatoplasty without complications or need for revision
* Non-CP cohort: have had prior adenoidectomy

Exclusion Criteria:

* Concurrent or past diagnosis of cancer or history of radiation
* Have or had vestibular pathology, cranial base surgery or ossicular chain reconstruction
* Craniofacial dysmorphology (other than non-syndromic CP with or without cleft lip in the CP cohort) or other syndrome
* A non-patent nasal cavity
* Patulous ET or pathologically low ET opening or closing pressures
* Unable or unwilling to perform the tests and exercises outlined in the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noel Jabbour, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) may be shared, after de-identification, with researchers who provide a methodologically sound proposal. IPD to be shared will include that necessary to achieve the aims in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 1 year after publication of summary data. Ending 5 years after publication.
Access Criteria: Proposals should be directed to shafferad@upmc.edu. To gain access, data requestors will need to sign data access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- EMST150: Subjects with or without cleft palate will use the EMST150 2 times a day for 8 weeks.
  EMST150: The EMST150 consists of a handheld plastic tube with a mouthpiece on one end and an adjustable valve on the other end. Your child will close his/her lips around the mouthpiece and breathe out against resistance. The EMST150 will be adjusted to the point where airflow stops. Each day, your child will blow into the EMST150 5 sets of 5 times with a 10-15 second rest between each use and a 1-2 minute rest between each set of 5. You will adjust the resistance of the device each week, take a picture of the device settings, and document exercise sets performed in an exercise diary. These exercises will be performed 2 times a day until your child's next visit at the MEPL (at least 8 weeks). Each session should take approximately 10-15 minutes, for a total of 30 minutes per day.
- EMST150 + Eustachi: Eustachi: The Eustachi has a handle attached to a nose probe that delivers a constant airflow into the nose. The Eustachi is turned on and while one nostril is pinched with one finger, the nose probe is sealed in the other nostril. Your child will swallow 5 times and will complete an exercise diary recording whether a popping or pressure change was felt in the left, right, or both ears. This exercise sequence will be performed twice in each nostril 2 times a day until your child's next visit at the MEPL (at least 8 weeks). Each session should take approximately 10-15 minutes, for a total of 30 minutes per day.
  EMST150: The EMST150 consists of a handheld plastic tube with a mouthpiece on one end and an adjustable valve on the other end. Your child will close his/her lips around the mouthpiece and breathe out against resistance. The EMST150 will be adjusted to the point where airflow stops. Each day, your child will blow into the EMST150 5 sets of 5 times with a 10-15 second rest between each use and a 1-2 minute rest between each set of 5. You will adjust the resistance of the device each week, take a picture of the device settings, and document exercise sets performed in an exercise diary. These exercises will be performed 2 times a day until your child's next visit at the MEPL (at least 8 weeks). Each session should take approximately 10-15 minutes, for a total of 30 minutes per day.
Period: Overall Study
Arm/Group | EMST150 | EMST150 + Eustachi
Started | 8 | 3
Visit 2 | 7 | 1
Visit 3 | 4 | 0
Completed | 4 | 0
Not Completed | 4 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — COVID-19 Restrictions | 1 | 2

BASELINE CHARACTERISTICS:
Population: For Eustachian Tube Function, analysis was performed on ears from which primary outcome data were available. Data were analyzed from 7 ears from 5 participants in the EMST150 group and 2 ears from 1 participant in the EMST150 + Eustachi group.
Units Other Than Participants: ears
Groups:
- EMST150: Subjects with or without cleft palate will use the EMST150 2 times a day for 8 weeks.
  The EMST150 consists of a handheld plastic tube with a mouthpiece on one end and an adjustable valve on the other end. Your child will close his/her lips around the mouthpiece and breathe out against resistance. The EMST150 will be adjusted to the point where airflow stops. Each day, your child will blow into the EMST150 5 sets of 5 times with a 10-15 second rest between each use and a 1-2 minute rest between each set of 5. You will adjust the resistance of the device each week, take a picture of the device settings, and document exercise sets performed in an exercise diary. These exercises will be performed 2 times a day until your child's next visit at the MEPL (at least 8 weeks). Each session should take approximately 10-15 minutes, for a total of 30 minutes per day.
- EMST150 + Eustachi: Subjects with or without cleft palate will use the EMST150 and Eustachi 2 times a day for 8 weeks.
  The Eustachi has a handle attached to a nose probe that delivers a constant airflow into the nose. The Eustachi is turned on and while one nostril is pinched with one finger, the nose probe is sealed in the other nostril. Your child will swallow 5 times and will complete an exercise diary recording whether a popping or pressure change was felt in the left, right, or both ears. This exercise sequence will be performed twice in each nostril 2 times a day until your child's next visit at the MEPL (at least 8 weeks). Each session should take approximately 10-15 minutes, for a total of 30 minutes per day.
  The EMST150 consists of a handheld plastic tube with a mouthpiece on one end and an adjustable valve on the other end. Your child will close his/her lips around the mouthpiece and breathe out against resistance. The EMST150 will be adjusted to the point where airflow stops. Each day, your child will blow into the EMST150 5 sets of 5 times with a 10-15 second rest between each use and a 1-2 minute rest between each set of 5. You will adjust the resistance of the device each week, take a picture of the device settings, and document exercise sets performed in an exercise diary. These exercises will be performed 2 times a day until your child's next visit at the MEPL (at least 8 weeks). Each session should take approximately 10-15 minutes, for a total of 30 minutes per day.
- Total: Total of all reporting groups
Arm/Group | EMST150 | EMST150 + Eustachi | Total
Number analyzed (Participants) | 8 | 3 | 11
Number analyzed (ears) | 7 | 2 | 9
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 10.9 [9.9 to 14.8] | 9.8 [9.7 to 15.2] | 10.6 [9.7 to 15.2]
Age, Customized [Count of Participants; unit: Participants]
  <10 years old | 2 | 2 | 4
  10-12 years old | 3 | 0 | 3
  >12 years old | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 3 | 10
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 3 | 10
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 3 | 11
Eustachian Tube Function [Median (Inter-Quartile Range); unit: percent change in middle ear pressure] — Percent change in middle ear pressure equilibrated during the inflation-deflation test at baseline Population: Eustachian tube function was analyzed for ears that had data for visit 2.
  percent change in middle ear pressure
    Inflation Test: number analyzed (Participants) | 5 | 1 | 6
    Inflation Test | 14.9 [9.6 to 50.8] | 81.2 [75.1 to 87.3] | 30.3 [14.8 to 67.5]
    Deflation Test | 5.7 [4.0 to 17.9] | 65.5 [30.5 to 100.5] | 10.7 [4.7 to 21.0]

OUTCOME MEASURES:

1. Primary Outcome: Eustachian Tube Function at 2 Months
Description: Percent change in middle ear pressure equilibrated during the inflation-deflation test at 2 months
Time Frame: 2 months
Population: In the EMST150 group, 2 participants were excluded because the inflation-deflation test was not able to be performed at visit 2 (due to patulous Eustachian tube or the ventilation tube being blocked). 1 participant was lost to follow-up. 3 ears with intact tympanic membranes from 3 participants were excluded
  2 participants in the EMST150 + Eustachi group were excluded from analysis. 1 was lost to follow-up after visit 1 and the other was unable to complete visit 2 prior to COVID restrictions.
Measure: Median (Inter-Quartile Range); unit: percent change in middle ear pressure
Units Other Than Participants: ears
Arm/Group | EMST150 | EMST150 + Eustachi
Number analyzed (Participants) | 5 | 1
Number analyzed (ears) | 7 | 2
percent change in middle ear pressure
  Inflation Test | 12.0 [10.4 to 65.8] | 83.6 [77.5 to 89.7]
  Deflation Test | 8.5 [4.7 to 10.4] | 44.0 [33.2 to 54.8]
Statistical Analysis 1: Comparison: EMST150; inflation test at 2 months compared with baseline; EMST150 + Eustachi not included because visit 2 measurements only available for 1 participant (2 ears); Test type: Other; p = 1.00, Wilcoxon signed-rank
Statistical Analysis 2: Comparison: EMST150; deflation test at 2 months compared with baseline; EMST150 + Eustachi not included because visit 2 measurements only available for 1 participant (2 ears); Test type: Other; p = 0.734, Wilcoxon signed-rank

2. Secondary Outcome: Eustachian Tube Function at 4 Months
Description: Percent change in middle ear pressure equilibrated during the inflation-deflation test at 4 months
Time Frame: 4 months
Population: 4 participants completed visit 3 (all in the EMST150 group). The inflation-deflation test was not completed in 2 participants because both tympanic membranes were intact. Of the 2 other participants, testing was able to be completed for both ears for 1. The other had testing completed in 1 ear. The other ear was not tested because the tympanic membrane was intact.
Measure: Median (Full Range); unit: percent change in middle ear pressure
Units Other Than Participants: ears
Arm/Group | EMST150
Number analyzed (Participants) | 2
Number analyzed (ears) | 3
percent change in middle ear pressure
  Inflation Test | 64.1 [23.0 to 87.2]
  Deflation Test | 6.5 [6.0 to 9.9]
Statistical Analysis 1: Comparison: EMST150; inflation test at 4 months compared with baseline; Test type: Other; p = 0.25, Wilcoxon signed-rank
Statistical Analysis 2: Comparison: EMST150; deflation test at 4 months compared with baseline; Test type: Other; p = 0.75, Wilcoxon signed-rank

3. Secondary Outcome: Eustachian Tube Function at 4 Months
Description: Percent change in middle ear pressure equilibrated during the inflation-deflation test at 4 months
Time Frame: 4 months
Population: as for outcome 2
Measure: Median (Full Range); unit: percent change in middle ear pressure
Units Other Than Participants: ears
Arm/Group | EMST150
Number analyzed (Participants) | 2
Number analyzed (ears) | 3
percent change in middle ear pressure
  Inflation Test | 64.1 [23.0 to 87.2]
  Deflation Test | 6.5 [6.0 to 9.9]
Statistical Analysis 1: Comparison: EMST150; inflation test at 4 months compared with 2 months; Test type: Other; p = 0.25, Wilcoxon signed-rank
Statistical Analysis 2: Comparison: EMST150; deflation test at 4 months compared with 2 months; Test type: Other; p = 0.75, Wilcoxon signed-rank

4. Other Pre Specified Outcome: Signs of Submucous Cleft Palate Following 2 Months of Exercise Compared With Baseline
Description: Presence or absence of dimpling anterior to the uvula, soft palate vaulting, midline groove, translucent midline, or visible notch in posterior hard palate observed on palate activation during video-analysis
Time Frame: Baseline and 2 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Signs of Submucous Cleft Palate Following 2 Months of Rest Compared With Baseline
Description: as for outcome 4
Time Frame: Baseline and 4 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Signs of Submucous Cleft Palate Following 2 Months of Rest Compared With Immediately Following 2 Months of Exercise
Description: as for outcome 4
Time Frame: 2 months and 4 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Perceptual Speech Symptoms of Velopharyngeal Dysfunction Following 2 Months of Exercise Compared With Baseline
Description: Perceptual symptoms of velopharyngeal incompetence measured using the Pittsburgh Weighted Speech Score, on a scale of 0-23, with ≥7 indicating likely velopharyngeal incompetence
Time Frame: Baseline and 2 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Perceptual Speech Symptoms of Velopharyngeal Dysfunction Following 2 Months of Rest Compared With Baseline
Description: as for outcome 7
Time Frame: Baseline and 4 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Perceptual Speech Symptoms of Velopharyngeal Dysfunction Following 2 Months of Rest Compared With Immediately Following 2 Months of Exercise
Description: as for outcome 7
Time Frame: 2 months and 4 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Eustachian Tube Function Observed During Maneuvers Following 2 Months of Exercise Compared With Baseline
Description: Maximum middle ear pressures achieved during Toynbee, Valsalva, Sniffing, Dive maneuver and the Patulous Test in daPa
Time Frame: Baseline and 2 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Residual Middle Ear Pressure Observed During Maneuvers Following 2 Months of Exercise Compared With Baseline
Description: Residual middle ear pressures achieved during Toynbee, Valsalva, Sniffing, Dive maneuver and the Patulous Test in daPa
Time Frame: Baseline and 2 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Eustachian Tube Function Observed During Maneuvers Following 2 Months of Rest Compared With Baseline
Description: Maximum middle ear pressures achieved during Toynbee, Valsalva, Sniffing, Dive maneuver and the Patulous Test in daPa
Time Frame: Baseline and 4 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Residual Middle Ear Pressure Observed During Maneuvers Following 2 Months of Rest Compared With Baseline
Description: Residual middle ear pressures achieved during Toynbee, Valsalva, Sniffing, Dive maneuver and the Patulous Test in daPa
Time Frame: Baseline and 4 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Eustachian Tube Function Observed During Maneuvers Following 2 Months of Rest Compared With Immediately Following 2 Months of Exercise
Description: Maximum middle ear pressures achieved during Toynbee, Valsalva, Sniffing, Dive maneuver and the Patulous Test in daPa
Time Frame: 2 months and 4 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Residual Middle Ear Pressure Observed During Maneuvers Following 2 Months of Rest Compared With Immediately Following 2 Months of Exercise
Description: Residual middle ear pressures achieved during Toynbee, Valsalva, Sniffing, Dive maneuver and the Patulous Test in daPa
Time Frame: 2 months and 4 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Velopharyngeal Function Observed During Maneuvers Following 2 Months of Exercise Compared With Baseline
Description: Maximum nasopharyngeal pressures achieved during Toynbee, Valsalva, Sniffing, Dive maneuver and the Patulous Test in daPa
Time Frame: Baseline and 2 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Residual Nasopharyngeal Pressures Observed During Maneuvers Following 2 Months of Exercise Compared With Baseline
Description: Residual nasopharyngeal pressures achieved during Toynbee, Valsalva, Sniffing, Dive maneuver and the Patulous Test in daPa
Time Frame: Baseline and 2 months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Velopharyngeal Function Observed During Maneuvers Following 2 Months of Rest Compared With Baseline
Description: as for outcome 16
Time Frame: Baseline and 4 months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Residual Nasopharyngeal Pressures Observed During Maneuvers Following 2 Months of Rest Compared With Baseline
Description: as for outcome 17
Time Frame: Baseline and 4 months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Velopharyngeal Function Observed During Maneuvers Following 2 Months of Rest Compared With Immediately Following 2 Months of Exercise
Description: as for outcome 16
Time Frame: 2 months and 4 months
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Residual Nasopharyngeal Pressures Observed During Maneuvers Following 2 Months of Rest Compared With Immediately Following 2 Months of Exercise
Description: as for outcome 17
Time Frame: 2 months and 4 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | EMST150 | EMST150 + Eustachi
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3
Other Adverse Events (participants affected / at risk) | 6/8 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EMST150 (N=8) | EMST150 + Eustachi (N=3)
Epistaxis (General disorders) | 1 (2) | 2 (2)
Otalgia (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Upper Respiratory Infection (General disorders) | 4 (4) | 3 (7)
Gastrointestinal Discomfort or Infection (General disorders) | 0 (0) | 2 (3)
Patulous Eustachian Tube (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Acute Otitis Media (Ear and labyrinth disorders) | 1 (1) | 0 (0)
COVID-19 (General disorders) | 1 (1) | 0 (0)
Allergic Rhinitis Symptoms (General disorders) | 1 (2) | 0 (0)
Bloody Otorrhea (Ear and labyrinth disorders) | 1 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment was limited due in part to delays related to COVID-19 restrictions. Another important limiting factor was the studied population itself. Inclusion/exclusion criteria were restrictive, and children who have persistent need for ventilation tubes frequently present with otorrhea or middle ear inflammation or tubes become blocked. These factors affect the feasibility of ETF tests and delayed study visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT03868891/Prot_SAP_000.pdf